CLINICAL TRIAL: NCT06692465
Title: A Multicenter, Randomized, Double-blind, Placebo -Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of GT20029 Solution in the Treatment of Androgenetic Alopecia (AGA) in Chinese Adult Males
Brief Title: To Evaluate the Efficacy and Safety of GT20029 Solution in the Treatment of Androgenetic Alopecia (AGA) in Chinese Adult Males
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Collaborators: Suzhou Koshine Biomedica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GT20029-CN-1002
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-06

CONDITIONS: Alopecia; Male Pattern Hair Loss
Keywords: Androgenetic Alopecia; Hair loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: GT20029 (Experimental)
  Interventions: Drug: GT20029 Tincture
- Placebo Comparator: GT20029 Matching Placebo (Placebo Comparator)
  Interventions: Drug: GT20029 matching placebo

INTERVENTIONS:
Drug: GT20029 Tincture — 5mg (0.5%) and 10mg (1%) one single dose per day (QD) treatment over 12 weeks period; 5mg (0.5%) and 10mg (1%) twice per week (BIW) treatment, on every Monday and Thursday over 12 weeks period
  Arms: Experimental: GT20029
Drug: GT20029 matching placebo — 5mg (0.5%) and 10mg (1%) matching placebo one single dose per day (QD) treatment over 12 weeks period; 5mg (0.5%) and 10mg (1%) matching placebo twice per week (BIW) treatment, on every Monday and Thursday over 12 weeks period
  Arms: Placebo Comparator: GT20029 Matching Placebo

SUMMARY:
The study is a multicenter, randomized, double-blind, placebo-controlled phase II clinical study to evaluate the efficacy and safety of GT20029 solution.

DETAILED DESCRIPTION:
GT20029 is a new investigational androgen receptor (AR) degrader for the treatment of androgenetic alopecia. A total of 180 adult male subjects with androgenetic alopecia (AGA) (according to Hamilton-Norwood classification IIIv, IV and V) were enrolled in this study. All subjects were randomly assigned in a 1:1:1:1:1:1ratio to investigational drug groups A, B, C and D and placebo groups E and F (i.e., 30 subjects in each group) and treated for 12 weeks at the specified dose and frequency for each group. The primary endpoint of the study is to evaluate the efficacy and safety of GT20029 solution in the treatment of androgenetic alopecia (AGA) in Chinese adult males and to determine the recommended dose for phase III trials.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the trial treatment plan and visit plan, voluntarily enroll, and sign the informed consent form in writing.
2. Male, aged ≥ 18 years old, in good overall health;
3. Clinical diagnosis of androgenetic alopecia (refer to 2019 edition of Chinese Guidelines for the Diagnosis and Treatment of Androgenetic Alopecia);
4. Alopecia severity according to Hamilton-Norwood classification IIIv, IV, V;
5. Willing to maintain the same hair style, hair color and hair length throughout the trial;
6. No parenting plan and able to use highly effective contraception during the trial and for 3 months after the last dose.

Exclusion Criteria:

1. History of severe systemic diseases/surgical history, which may affect the safety and efficacy evaluation of the investigational drug, such as circulatory system, nervous system, blood system, digestive system (such as inflammatory bowel disease), immune system, mental system diseases;
2. Alopecia areata or diffuse alopecia areata, syphilis alopecia, cicatricial alopecia, malnutrition, chemotherapy/radiotherapy caused by alopecia;
3. Patients with scalp skin diseases that affect the efficacy evaluation, trauma in the target area of the scalp or other scalp skin lesions requiring topical drug treatment, such as fungal or bacterial infections, severe seborrheic dermatitis, scalp psoriasis, contact dermatitis, severe folliculitis or scalp atrophy;
4. Combined with diseases that have an impact on hair growth, such as connective tissue disease, moderate to severe anemia, and significant weight loss in a short period of time;
5. Patients who have a history of hair transplantation or need to wear wig hair cover for a long time during the trial treatment;
6. Combined with endocrine related diseases affecting androgen levels, including but not limited to male testicular disease, Klinefelter syndrome, diseases affecting the hypothalamus-pituitary-gonadal axis;
7. Use of Chinese patent medicine drugs, food and health products with alopecia treatment 1 month before screening, such as Yangxue Shengfa Capsules, Lingdan Tablets, Zhangguang 101 germinal fluid, and Caifei Germinative fluid;
8. Patients who have taken androgen replacement therapy, immunosuppressive agents, corticosteroids preparations and other drugs that may interfere with the efficacy evaluation within 3 months before screening;
9. Use of minoxidil within 6 months before screening;
10. Patients treated with oral finasteride or dutasteride within 12 months before screening;
11. Patients who have used topical drugs for alopecia sites within 3 months before screening;
12. Receiving scalp radiation and/or laser or surgical therapy within 3 months before screening;
13. Use of other medical shampoos or solutions containing ketoconazole or similar ingredients (eg. Terzolin) that may interfere with the efficacy evaluation within 1 month before screening;
14. Allergic to the investigational drug or known to be allergic to the ingredients of the study product;
15. Abnormal and clinically significant physical examination, vital signs, 12-lead ECG, blood routine, urine routine, blood biochemistry, sex hormone tests during the screening period, and judged by the investigator to affect the efficacy and safety evaluation of subjects and test results;
16. Any or more of the results of human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen or hepatitis C virus antibody are positive;
17. Participating or participating in ongoing interventional drug or medical device clinical trials within 3 months before screening;
18. History of drug abuse within 1 year before screening;
19. Consumption of more than 14 units of alcohol per week (1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine) within 3 months before screening;
20. Major surgery within 3 months before screening, or plan to undergo major surgery during the trial;
21. Other conditions that may affect compliance or unsuitable for participating in this study in the investigator 's opinion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in non-vellus hair count (TAHC, Target Area Hair Counts) within target area (change from baseline at 12 weeks of treatment) | 12 weeks
  Changes from baseline in non-vellus TAHC (Target Area Hair Counts) (Non-vellus TAHC is the number of non-vellus hairs within 1 cm² scalp, which usually ranges from 0 to 300. Larger non-vellus TAHC implies thicker hair. In this study, larger change in non-vellus TAHC means better outcome.)

SECONDARY OUTCOMES:
Hair growth (HGA) assessment, including subject self-assessment and investigator assessment (change from baseline at 6 and 12 weeks of treatment) | 6 weeks, 12 weeks
  Changes from baseline HGA (Hair Growth Assessment) score by Principal Investigator and subjects (HGA scale ranged from -3 to 3 and represented decreases from baseline that were substantial, moderate, slight, no change, slight increases, moderate increases, and substantial increases, respectively. HGA improvement was defined as a hair growth assessment score of larger than 0.)
TAHC assessment | 6 weeks
  Change in non-vellus hair count (TAHC) in the target area (change from baseline at 6 weeks of treatment)
TAHW assessment | 6 weeks, 12 weeks
  Change in non-vellus hair diameter (TAHW) in the target area (change from baseline at 6 and 12 weeks of treatment)
Terminal hair/vellus hair ratio assessment | 6 weeks, 12 weeks
  Change in terminal hair/vellus hair ratio (change from baseline at 6 and 12 weeks of treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology department, Huashan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No